CLINICAL TRIAL: NCT02737605
Title: A Randomized, Double-Blind (Periods 1 to 3), Placebo- and Positive-Controlled, Single Dose, 4-Period, Crossover Study to Evaluate the Effects of Esketamine on Cardiac Repolarization in Healthy Subjects
Brief Title: A Study to Evaluate the Effects of Esketamine on Cardiac Repolarization in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR106218; 2014-004457-14 (EudraCT Number); ESKETINTRD1013 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-04-08; First posted 2016-04-14 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Healthy
Keywords: Esketamine; Healthy; Pharmacokinetics; Electrocardiogram; Repolarization
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (6):
- Sequence 1 (Experimental): Participants will receive Treatment A (intravenous placebo, Intranasal placebo and Oral placebo tablet matched to the moxifloxacin tablet) on Day 1 of period 1, Treatment B (intravenous placebo, 84 milligram (mg) of intranasal esketamine and Oral placebo tablet matched to the moxifloxacin tablet) on Day 1 of period 2, Treatment C (intravenous placebo, Intranasal placebo and 400 mg oral moxifloxacin tablet) on Day 1 of period 3, Treatment D (0.8 milligram per kilogram of intravenous esketamine, Intranasal placebo and Oral placebo tablet matched to the moxifloxacin tablet ) on Day 1 of period 4. Periods 1, 2, 3 and 4 will be separated by 5 to 7 days.
  Interventions: Drug: Intranasal Esketamine; Drug: Intravenous Esketamine; Drug: Moxifloxacin; Drug: Oral Placebo; Drug: Intravenous Placebo; Drug: Intranasal Placebo
- Sequence 2 (Experimental): Participants will receive Treatment A on Day 1 of period 1, Treatment C on Day 1 of period 2, Treatment B on Day 1 of period 3, Treatment D on Day 1 of period 4. Periods 1, 2, 3 and 4 will be separated by 5 to 7 days.
  Interventions: Drug: Intranasal Esketamine; Drug: Intravenous Esketamine; Drug: Moxifloxacin; Drug: Oral Placebo; Drug: Intravenous Placebo; Drug: Intranasal Placebo
- Sequence 3 (Experimental): Participants will receive Treatment B on Day 1 of period 1, Treatment C on Day 1 of period 2, Treatment A on Day 1 of period 3, Treatment D on Day 1 of period 4. Periods 1, 2, 3 and 4 will be separated by 5 to 7 days.
  Interventions: Drug: Intranasal Esketamine; Drug: Intravenous Esketamine; Drug: Moxifloxacin; Drug: Oral Placebo; Drug: Intravenous Placebo; Drug: Intranasal Placebo
- Sequence 4 (Experimental): Participants will receive Treatment B on Day 1 of period 1, Treatment A on Day 1 of period 2, Treatment C on Day 1 of period 3, Treatment D on Day 1 of period 4. Periods 1, 2, 3 and 4 will be separated by 5 to 7 days.
  Interventions: Drug: Intranasal Esketamine; Drug: Intravenous Esketamine; Drug: Moxifloxacin; Drug: Oral Placebo; Drug: Intravenous Placebo; Drug: Intranasal Placebo
- Sequence 5 (Experimental): Participants will receive Treatment C on Day 1 of period 1, Treatment A on Day 1 of period 2, Treatment B on Day 1 of period 3, Treatment D on Day 1 of period 4. Periods 1, 2, 3 and 4 will be separated by 5 to 7 days.
  Interventions: Drug: Intranasal Esketamine; Drug: Intravenous Esketamine; Drug: Moxifloxacin; Drug: Oral Placebo; Drug: Intravenous Placebo; Drug: Intranasal Placebo
- Sequence 6 (Experimental): Participants will receive Treatment C on Day 1 of period 1, Treatment B on Day 1 of period 2, Treatment A on Day 1 of period 3, Treatment D on Day 1 of period 4. Periods 1, 2, 3 and 4 will be separated by 5 to 7 days.
  Interventions: Drug: Intranasal Esketamine; Drug: Intravenous Esketamine; Drug: Moxifloxacin; Drug: Oral Placebo; Drug: Intravenous Placebo; Drug: Intranasal Placebo

INTERVENTIONS:
Drug: Intranasal Esketamine — Participants will receive 84 mg intranasal esketamine as 3 devices, each with 28 mg esketamine.
Drug: Intravenous Esketamine — Participants will receive 0.8 milligram per kilogram body weight esketamine, 40 minutes, intravenous infusion.
Drug: Moxifloxacin — Participants will receive 400 mg Moxifloxacin orally.
Drug: Oral Placebo — Participants will receive matching placebo orally.
Drug: Intravenous Placebo — Participants will receive placebo 40 minutes, intravenous infusion.
Drug: Intranasal Placebo — Participants will receive intranasal placebo (1 spray in each nostril at 0, 5, and 10 minutes).

SUMMARY:
The purpose of the study is to assess the effects of esketamine on QT/QTc intervals and electrocardiogram (ECG) morphology at therapeutic exposures of esketamine and noresketamine (intranasal administration) and supratherapeutic exposures of esketamine (intravenous administration) in healthy adults.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned to participants by chance), placebo- and positive-controlled, double-blind (Periods 1 to 3), and open-label (Period 4), single-dose, crossover study in up to 60 healthy adults. The study has a Screening Phase and a Treatment Phase. Participants will be randomly assigned to 1 of 6 treatment sequence groups and will receive the 4 treatments (1 treatment per period); Treatment A (intravenous placebo, Intranasal placebo and Oral placebo tablet matched to the moxifloxacin tablet), Treatment B (intravenous placebo, 84 milligram (mg) of intranasal esketamine as 4 devices, each with 28 mg esketamine and Oral placebo tablet matched to the moxifloxacin tablet), Treatment C (intravenous placebo, Intranasal placebo and 400 mg oral moxifloxacin tablet) and Treatment D (0.8 milligram per kilogram of intravenous esketamine, Intranasal placebo and Oral placebo tablet matched to the moxifloxacin tablet ). The first 3 periods will be double-blinded and the fourth period will be open-label. Periods 1, 2, 3, and 4 will be separated by 5 to 7 days. Primarily the effects of esketamine on QT/QTc intervals and electrocardiogram (ECG) morphology will be evaluated. Safety of the participants will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* Body mass index (BMI) between 18 and 30 kilogram (kg)/meter square ([m]^2) (inclusive), and body weight not less than 50 kilogram (kg)
* Women using oral contraceptives must agree to use an additional birth control method during the study and for 1 month after receiving the last dose of study drug or until after the next menstrual period
* A woman of child-bearing potential, must have a negative serum beta-human chorionic gonadotropin (hCG) pregnancy test at Screening and a negative urine pregnancy test on Day -1 of the first treatment period
* A man, must agree to use an adequate contraception method as deemed appropriate by the investigator (example, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Participant has a current diagnosis of psychotic disorder or major depressive disorder (MDD) with psychosis, bipolar or related disorders, intellectual disability, borderline personality disorder, or antisocial personality disorder
* Clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, gastrointestinal disease, hypertension, vascular disorders, sleep apnea, myasthenia gravis, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* History of additional risk factors for torsade de pointes or the presence of a family history of Short QT Syndrome, Long QT Syndrome, sudden unexplained death at a young age (less than/equal to 40 years), drowning or sudden infant death syndrome in a first degree relative (that is, biological parent, sibling, or child)
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at Screening or at admission to the study center for the first treatment period as deemed appropriate by the investigator. Electrolytes (potassium, magnesium, calcium) should be within the reference range of the laboratory
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) at Screening or at admission to the study center for the first treatment period as deemed appropriate by the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Mean Change From Baseline in QTc Interval | Up to Day 2
  The QT interval corrected for heart rate (QTc interval) using Fridericia, Bazett and study-specific power correction methods, will be measured by electrocardiograms (ECG).
Percentage of Participants With Maximum Change From Baseline in Electrocardiogram (ECG) Morphology | Up to Day 2

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Predose, 0.25, 0.33, 0.5, 0.67, 0.83, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24 and 30 hours post-dose on Day 1
  Cmax is defined as maximum observed analyte concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Predose, 0.25, 0.33, 0.5, 0.67, 0.83, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24 and 30 hours post-dose on Day 1
  Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration Time Curve From Time Zero to 12 Hours (AUC [0-12]) | Predose, 0.25, 0.33, 0.5, 0.67, 0.83, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24 and 30 hours post-dose on Day 1
  The AUC (0-12) is the area under the plasma concentration time curve from time 0 to 12 hours post-dose.
Area Under the Plasma Concentration Time Curve From Time Zero to Time at Last Observed Quantifiable Concentration (AUClast) | Predose, 0.25, 0.33, 0.5, 0.67, 0.83, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24 and 30 hours post-dose on Day 1
  The AUClast is area under the plasma concentration time curve from time zero to the last quantifiable concentration.
Area Under the Plasma Concentration Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Predose, 0.25, 0.33, 0.5, 0.67, 0.83, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24 and 30 hours post-dose on Day 1
  The AUC (0-infinity) is area under the plasma concentration time curve from time zero to infinite time, calculated as the sum of Area under Curve (AUC) last and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration.
Elimination Half-life Period (T1/2) | Predose, 0.25, 0.33, 0.5, 0.67, 0.83, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24 and 30 hours post-dose on Day 1
  T1/2 is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal rate-constant (lambda[z]) of the semi logarithmic drug concentrationtime curve, and is calculated as 0.693/lambda(z).
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Screening to follow-up visit (within 10 plus or minus 2 days after last dose administration)
Change From Baseline in Heart rate | Up to Day 2
Change From Baseline in QRS Interval | Up to Day 2
Change From Baseline in PR Interval | Up to Day 2
Change From Baseline in RR Interval | Up to Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Berlin, Germany